CLINICAL TRIAL: NCT06107257
Title: Cardiogenic Acute Pulmonary Edema in Subjects Over 75 Years Old: Impact of Non-invasive Ventilation on Mortality
Acronym: CAPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8785
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Cardiogenic Pulmonary Edema
Keywords: Cardiogenic Pulmonary Edema; Acute pulmonary edema; Non-invasive ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People aged over 75 represent almost 10% of the general population, and 12 to 14% of patients consulting emergency departments. Cardiogenic acute pulmonary edema (APO) is a very common reason for admission to the emergency room. The effectiveness of non-invasive ventilation (NIV) has been demonstrated during the management of PAO and would allow, compared to medical treatment alone, a more rapid improvement in clinical and gasometric parameters as well as a reduction in the need for ventilation. orotracheal intubation. On the other hand, the impact of NIV on mortality in cardiogenic PAO seems poorly defined, with lower levels of scientific evidence regarding a possible benefit in terms of survival, particularly in the elderly population.

The objective of this study is to determine whether the use of NIV in cardiogenic PAO in elderly subjects admitted to the emergency room of Strasbourg University Hospital would have an impact in terms of mortality up to 6 months compared to medical treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (> 75 years old)
* Admission to the NHC emergency room between January 1, 2021 and October 31, 2021
* Diagnosis of cardiogenic PAO
* Indication of NIV according to current recommendations
* Subject not opposing the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his opposition to the reuse of his data for scientific research purposes.
* Presence of an absolute contraindication to NIV
* Respiratory distress due to pneumonia or other diagnosis
* RT-PCR Sars Cov 2 positive in emergency

Min Age: 76 Years | Sex: All
Age Groups: Older Adult
Study Population: Adult subject (> 75 years) with a diagnosis of cardiogenic PAO treated at Strasbourg University Hospital between January 1, 2021 and October 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival Analysis | 6 months after cardiogenic acute pulmonary edema

CONTACTS AND LOCATIONS:
Locations (1):
- Gériatrie - Service de Soins de Soins Médicaux et de Réadaptation - CHU de Strasbourg - France, Strasbourg, France

REFERENCES:
- [Derived] Haddi L, Valerio L, Bilbault P, Kaltenbach G, Schmitt E. Effect of noninvasive ventilation on 6-month mortality in patients with acute cardiogenic pulmonary oedema: a retrospective study dedicated to older persons. Intern Emerg Med. 2025 Sep;20(6):1753-1760. doi: 10.1007/s11739-025-04012-3. Epub 2025 Jun 15. PMID 40517332